CLINICAL TRIAL: NCT04294576
Title: First-in-human (FIH), Open-Label, Phase 1a (Dose Escalation)/Phase 1b (Expansion Cohort) Trial of BJ-001 as a Single Agent and in Combination With Pembrolizumab in Patients With Locally Advanced/Metastatic Solid Tumors
Brief Title: Safety Study of BJ-001, an IL-15 Fusion Protein, for Locally Advanced/Metastatic Solid Tumors
Acronym: FIH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BJ Bioscience, Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BJ-001-01-001US; KEYNOTE-F13 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-02-07; First posted 2020-03-04 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced/Metastatic Solid Tumors
Keywords: FIH; Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Masking Description: no masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1; BJ-001 (Experimental): Phase 1a Part 1, Part 2, and Part 4: dose escalation for BJ-001 as single agent
  Interventions: Drug: BJ-001
- Arm 2; BJ-001 and pembrolizumab (Experimental): Phase 1a Part 3 and Part 5: dose escalation for BJ-001 in combination with Pembrolizumab
  Phase 1b: expansion cohorts for the combination of BJ-001 and pembrolizumab
  Interventions: Drug: BJ-001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BJ-001 — BJ-001 dosed via SC injection as single agent. One cycle is 6 weeks.
Drug: Pembrolizumab — BJ-001 dosed via SC injection in combination with Pembrolizumab
  One cycle is 6 weeks.
  Other Names: Keytruda
  Arms: Arm 2; BJ-001 and pembrolizumab

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BJ-001, a human IL-15 fusion protein, administered via subcutaneous injections, as a single agent and in combination with pembrolizumab in adult patients with Locally Advanced/Metastatic Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a patients must have locally advanced or metastatic solid tumors,
* Phase 1b patients must have locally advanced or metastatic and/or non-resectable head and neck squamous cell carcinoma, cholangiocarcinoma, stomach cancer, melanoma, pancreatic cancer, NSCLC (as high expression of αVβ3, αVβ5, or αVβ6 have been reported for these tumors)

  * Measurable disease: For Phase 1a patients can have non-measurable or measurable disease. For all other parts: measurable disease defined by RECIST v1.1 is required
  * For Phase 1a Part 3 and Phase 1b patients (combination treatment) must be refractory or relapsed to anti-PD-1, anti-PD-L1 or anti-CTLA4 checkpoint inhibitors for all tumor types, For Part 1 and Part 2 of Phase 1a (BJ-001 single agent treatment) both checkpoint inhibitor naïve or refractory/relapsed patients will be considered.
* Patient who have diagnosis for which treatment with pembrolizumab to be enrolled. Patients previously treated with pembrolizumab and who have progressed are eligible. to be enrolled.

  * Adequate hematologic function,
  * Adequate hepatic function, defined by all of the following:
  * Adequate renal function defined by estimated creatinine clearance ≥ 45 mL/min (Cockcroft and Gault formula
  * ECOG Performance Status (PS) of 0-2.
  * No history of any hematopoietic malignancy.
  * No active or history of clinically significant autoimmune disease (as defined by previously requiring immunosuppressive therapy).

Exclusion Criteria:

* Pregnant or nursing females.
* Receipt of any investigational product or any approved anticancer drug(s) or biological product(s) within 4 weeks prior to the first dose of study drug. Exceptions: Hormone replacement therapy, testosterone, or oral contraceptives (LHRH antagonists are allowed).
* Patients previously treated with an anti PD-1/PD-L1 targeting agent who have had any prior history of immune-mediated pneumonitis, any immune-mediated toxicity of ≥ Grade 3,
* Patients with a history of severe allergic or anaphylactic reactions to human mAb therapy or known hypersensitivity.
* Patients with a history of pneumonitis, myocarditis, history of Stevens-Johnson syndrome or toxic epidermal necrolysis.
* Patients who have undergone a bone marrow transplantation, solid organ transplantation, or stem cell transplant.
* Patients with unresolved AEs > Grade 1 from prior anticancer therapy.
* Patients who have received prior interferon or IL-2 therapy less than 4 weeks prior to enrollment.
* Uncontrolled primary central nervous system (CNS) tumors or CNS metastases; based on screening.
* Patients with active autoimmune disease or a documented medical history of autoimmune disease managed by replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2024-04-29 (Estimated); Study Completion 2024-10-22 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAE | 90 days after the last dose
  To assess the safety and tolerability of BJ-001 as a single agent administered s.c. at escalating dose levels in adults with solid tumors.
Severity of AEs in patients with solid tumors enrolled in the study. | From Day 1 of treatment up to 30 days after last dose
  To assess the safety and tolerability of s.c. BJ-001 administered at escalating dose levels in combination with Pembrolizumab inhibitor. in adults with solid tumors.
Dose limiting toxicities (DLTs) BJ-001 as a single agent | at the end of week 4 after first dose
  To determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of BJ-001 as a single agent.
Dose limiting toxicities (DLTs) BJ-001 in combination with pembrolizumab inhibitor. | at the end of week 4 after first dose
  To determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of s.c. BJ-001 administered at escalating dose levels in combination with pembrolizumab in adults with solid tumors.

SECONDARY OUTCOMES:
Immunogenicity of BJ-001 as a single agent and in combination with Pembrolizumab. | 90 days after last dose
  The frequency of anti-drug antibodies (ADA) against BJ-001 as a single agent and in combination with Pembrolizumab.
Pharmacokinetic (PK) AUC0-τ samples patients treated with BJ-001 as a single agent and in combination with Pembrolizumab. | 24 weeks
  PK parameters (AUC0-τ) following the first dose and the fourth dose
Pharmacokinetic (PK) Cmax samples patients treated with BJ-001 as a single agent and in combination with Pembrolizumab. | 24 weeks
  PK parameters (Cmax) following the first dose and the fourth dose
Pharmacokinetic (PK) Ctrough samples patients treated with BJ-001 as a single agent and in combination with Pembrolizumab. | 24 weeks
  PK parameters (Ctrough) following the first dose and the fourth dose
Pharmacokinetic (PK) Tmax samples patients treated with BJ-001 as a single agent and in combination with Pembrolizumab. | 24 weeks
  PK parameters (Tmax) following the first dose and the fourth dose

CONTACTS AND LOCATIONS:
Overall Officials: Joe Zhang, PhD, Study Director — BJ Bioscience
Locations (5):
- United States (5):
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai, New York, New York
  - Greenville Hospital System University Medical Center (ITOR), Greenville, South Carolina
  - NEXT Oncology, San Antonio, Texas
  - Northwest Medical Specialities, Tacoma, Washington

REFERENCES:
- [Background] Brahmer JR, Lacchetti C, Schneider BJ, Atkins MB, Brassil KJ, Caterino JM, Chau I, Ernstoff MS, Gardner JM, Ginex P, Hallmeyer S, Holter Chakrabarty J, Leighl NB, Mammen JS, McDermott DF, Naing A, Nastoupil LJ, Phillips T, Porter LD, Puzanov I, Reichner CA, Santomasso BD, Seigel C, Spira A, Suarez-Almazor ME, Wang Y, Weber JS, Wolchok JD, Thompson JA; National Comprehensive Cancer Network. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2018 Jun 10;36(17):1714-1768. doi: 10.1200/JCO.2017.77.6385. Epub 2018 Feb 14. PMID 29442540
- [Background] Caudana P, Nunez NG, De La Rochere P, Pinto A, Denizeau J, Alonso R, Niborski LL, Lantz O, Sedlik C, Piaggio E. IL2/Anti-IL2 Complex Combined with CTLA-4, But Not PD-1, Blockade Rescues Antitumor NK Cell Function by Regulatory T-cell Modulation. Cancer Immunol Res. 2019 Mar;7(3):443-457. doi: 10.1158/2326-6066.CIR-18-0697. Epub 2019 Jan 16. PMID 30651291
- [Background] Conlon KC, Lugli E, Welles HC, Rosenberg SA, Fojo AT, Morris JC, Fleisher TA, Dubois SP, Perera LP, Stewart DM, Goldman CK, Bryant BR, Decker JM, Chen J, Worthy TA, Figg WD Sr, Peer CJ, Sneller MC, Lane HC, Yovandich JL, Creekmore SP, Roederer M, Waldmann TA. Redistribution, hyperproliferation, activation of natural killer cells and CD8 T cells, and cytokine production during first-in-human clinical trial of recombinant human interleukin-15 in patients with cancer. J Clin Oncol. 2015 Jan 1;33(1):74-82. doi: 10.1200/JCO.2014.57.3329. Epub 2014 Nov 17. PMID 25403209
- [Background] Cox L, Larenas-Linnemann D, Lockey RF, Passalacqua G. Speaking the same language: The World Allergy Organization Subcutaneous Immunotherapy Systemic Reaction Grading System. J Allergy Clin Immunol. 2010 Mar;125(3):569-74, 574.e1-574.e7. doi: 10.1016/j.jaci.2009.10.060. Epub 2010 Feb 7. PMID 20144472
- [Background] Desbois M, Le Vu P, Coutzac C, Marcheteau E, Beal C, Terme M, Gey A, Morisseau S, Teppaz G, Boselli L, Jacques Y, Bechard D, Tartour E, Cassard L, Chaput N. IL-15 Trans-Signaling with the Superagonist RLI Promotes Effector/Memory CD8+ T Cell Responses and Enhances Antitumor Activity of PD-1 Antagonists. J Immunol. 2016 Jul 1;197(1):168-78. doi: 10.4049/jimmunol.1600019. Epub 2016 May 23. PMID 27217584
- [Background] Hensley TR, Easter AB, Gerdts SE, De Rosa SC, Heit A, McElrath MJ, Andersen-Nissen E. Enumeration of major peripheral blood leukocyte populations for multicenter clinical trials using a whole blood phenotyping assay. J Vis Exp. 2012 Sep 16;(67):e4302. doi: 10.3791/4302. PMID 23007739
- [Background] Knudson KM, Hicks KC, Alter S, Schlom J, Gameiro SR. Mechanisms involved in IL-15 superagonist enhancement of anti-PD-L1 therapy. J Immunother Cancer. 2019 Mar 21;7(1):82. doi: 10.1186/s40425-019-0551-y. PMID 30898149
- [Background] Erratum: Lee DW, Gardner R, Porter DL, et al. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014;124(2):188-195. Blood. 2016 Sep 15;128(11):1533. doi: 10.1182/blood-2016-07-730689. PMID 31265503
- [Background] Lenz HJ. Management and preparedness for infusion and hypersensitivity reactions. Oncologist. 2007 May;12(5):601-9. doi: 10.1634/theoncologist.12-5-601. PMID 17522249
- [Background] Mier JW, Brandon EP, Libby P, Janicka MW, Aronson FR. Activated endothelial cells resist lymphokine-activated killer cell-mediated injury. Possible role of induced cytokines in limiting capillary leak during IL-2 therapy. J Immunol. 1989 Oct 1;143(7):2407-14. PMID 2528594
- [Background] Raedler LA. Opdivo (Nivolumab): Second PD-1 Inhibitor Receives FDA Approval for Unresectable or Metastatic Melanoma. Am Health Drug Benefits. 2015 Mar;8(Spec Feature):180-3. No abstract available. PMID 26629287
- [Background] Rhode PR, Egan JO, Xu W, Hong H, Webb GM, Chen X, Liu B, Zhu X, Wen J, You L, Kong L, Edwards AC, Han K, Shi S, Alter S, Sacha JB, Jeng EK, Cai W, Wong HC. Comparison of the Superagonist Complex, ALT-803, to IL15 as Cancer Immunotherapeutics in Animal Models. Cancer Immunol Res. 2016 Jan;4(1):49-60. doi: 10.1158/2326-6066.CIR-15-0093-T. Epub 2015 Oct 28. PMID 26511282
- [Background] Rosenberg SA. IL-2: the first effective immunotherapy for human cancer. J Immunol. 2014 Jun 15;192(12):5451-8. doi: 10.4049/jimmunol.1490019. PMID 24907378
- [Background] Sim GC, Radvanyi L. The IL-2 cytokine family in cancer immunotherapy. Cytokine Growth Factor Rev. 2014 Aug;25(4):377-90. doi: 10.1016/j.cytogfr.2014.07.018. Epub 2014 Aug 1. PMID 25200249
- [Background] Salmaninejad A, Valilou SF, Shabgah AG, Aslani S, Alimardani M, Pasdar A, Sahebkar A. PD-1/PD-L1 pathway: Basic biology and role in cancer immunotherapy. J Cell Physiol. 2019 Aug;234(10):16824-16837. doi: 10.1002/jcp.28358. Epub 2019 Feb 19. PMID 30784085
- [Background] Waldmann TA. The biology of interleukin-2 and interleukin-15: implications for cancer therapy and vaccine design. Nat Rev Immunol. 2006 Aug;6(8):595-601. doi: 10.1038/nri1901. PMID 16868550
- [Background] West EE, Jin HT, Rasheed AU, Penaloza-Macmaster P, Ha SJ, Tan WG, Youngblood B, Freeman GJ, Smith KA, Ahmed R. PD-L1 blockade synergizes with IL-2 therapy in reinvigorating exhausted T cells. J Clin Invest. 2013 Jun;123(6):2604-15. doi: 10.1172/JCI67008. Epub 2013 May 15. PMID 23676462
- [Background] Wrangle JM, Velcheti V, Patel MR, Garrett-Mayer E, Hill EG, Ravenel JG, Miller JS, Farhad M, Anderton K, Lindsey K, Taffaro-Neskey M, Sherman C, Suriano S, Swiderska-Syn M, Sion A, Harris J, Edwards AR, Rytlewski JA, Sanders CM, Yusko EC, Robinson MD, Krieg C, Redmond WL, Egan JO, Rhode PR, Jeng EK, Rock AD, Wong HC, Rubinstein MP. ALT-803, an IL-15 superagonist, in combination with nivolumab in patients with metastatic non-small cell lung cancer: a non-randomised, open-label, phase 1b trial. Lancet Oncol. 2018 May;19(5):694-704. doi: 10.1016/S1470-2045(18)30148-7. Epub 2018 Apr 5. PMID 29628312
- See also: KEYTRUDA (pembrolizumab), [package insert]. Merck Sharp & Dohme Corp. Whitehouse Station, NJ.2014. Accessed at Drugs@FDA: FDA Approved Drug Products on December 28, 2018. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125514s037lbl.pdf
- See also: OPDIVO (nivolumab), [package insert]. Bristol-Myers Squibb Company, Princeton, NJ. 2014. Accessed at Drugs@FDA: FDA Approved Drug Products on November 15, 2018. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125554s069lbl.pdf
- See also: TECENTRIQ (atezolizumab), [package insert]. Genentech, Inc. San Francisco, CA. 2016. Accessed at Drugs@FDA: FDA Approved Drug Products on December 6, 2018. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/761034s009lbl.pdf
- See also: YERVOY (ipilimumab), [package insert]. Bristol-Myers Squibb Company, Princeton, NJ. 2011. Accessed at Drugs@FDA: FDA Approved Drug Products on July 10, 2018. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125377s096lbl.pdf